CLINICAL TRIAL: NCT01353651
Title: Endovascular Versus Open Repair of the Common Femoral Artery: a Randomized Trial (TECCO)
Brief Title: Endovascular Versus Open Repair of the Common Femoral Artery
Acronym: TECCO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/6-Q
Record Dates: First submitted 2011-05-09; First posted 2011-05-13 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Atherosclerotic Lesions of the Common Femoral Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endovascular treatment (Experimental)
  Interventions: Device: Endovascular treatment using self expandable nitinol STENTS
- Open repair treatment (Active Comparator)
  Interventions: Device: Open repair treatment

INTERVENTIONS:
Device: Endovascular treatment using self expandable nitinol STENTS — A direct stenting will be performed.
  Arms: Endovascular treatment
Device: Open repair treatment — The surgeon will perform its usual technique to revascularize the common femoral artery
  Arms: Open repair treatment

SUMMARY:
Even though the indication for endovascular therapy has been enlarged, open repair of common femoral artery is still considered as the treatment of choice. A recent pilot study showed that endovascular repair of the CFA seems to be a safe technique of revascularization with acceptable initial results at 12 months (Azema et al, Eur J Vasc Endovasc Surg, 2011, in press). TECCO, a French randomized and controlled trial, has been set up to compare open and endovascular procedures for the treatment of CFA atherosclerotic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 90 years-old
* De novo atheromatous common femoral artery stenosis
* Symptomatic lesions (Rutherford stages 3, 4, 5 and 6)
* Haemodynamically significant lesion
* Written informed consent

Exclusion Criteria:

* Restenosis
* Non-atheromatous lesions (dysplasia, post-traumatic, inflammatory)
* external iliac thrombosis and / or common femoral side to treat
* Contraindication to open surgery or endovascular treatment
* Contraindication to anesthesia
* Indication of aorto-femoral, ilio-femoral, femoral-popliteal or femoro-tibialis bypass to associate with the common femoral revascularization
* Indication of a surgical approach to the external iliac artery through a retroperitoneal
* Asymptomatic lesions
* Life expectancy less than one year
* Refusing patient
* Inability to monitor during the test period
* Participation in another clinical trial
* Pregnant Women
* No written informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Morbid-mortality rate at 30 days | 30 days
  Morbid-mortality rate is defined by: Death, general complications and local complications requiring re-admission and / or reoperation.

SECONDARY OUTCOMES:
Technical success | 1 month
Hospital length of stay | 1 month
Primary sustained clinical improvement | 1 month
Primary sustained clinical improvement | 6 months
Primary sustained clinical improvement | 12 months
Primary sustained clinical improvement | 24 months
Target lesion revascularization | 1 month
Target lesion revascularization | 6 months
Target lesion revascularization | 12 months
Target lesion revascularization | 24 months
In-stent restenosis | 1 month
In-stent restenosis | 6 months
In-stent restenosis | 12 months
In-stent restenosis | 24 months
Stent fracture | 1 month
Stent fracture | 6 months
Stent fracture | 12 months
Stent fracture | 24 months
Secondary sustained clinical improvement | 1 month
Secondary sustained clinical improvement | 6 months
Secondary sustained clinical improvement | 12 months
Secondary sustained clinical improvement | 24 months
Target extremity revascularization | 1 month
Target extremity revascularization | 6 months
Target extremity revascularization | 12 months
Target extremity revascularization | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yann GOUEFFIC, Doctor, Principal Investigator — Nantes University Hospital
Locations (17):
- France (17):
  - University Hospital, Amiens
  - University Hospital, Besançon
  - University Hospital, Bordeaux
  - University Hospital, Clermont-Ferrand
  - University Hospital, Dijon
  - University Hospital, Lyon
  - University Hospital, Marseille
  - NCN Clinic, Nantes
  - St Augustin Clinic, Nantes
  - University Hospital, Nantes
  - University Hospital, Nice
  - University Hospital, HEGP, Paris
  - University Hospital, Henri Mondor, Paris
  - University Hospital, Rouen
  - University Hospital, Saint-Etienne
  - University Hospital, Strasbourg
  - Tonkin Clinic, Villeurbanne

REFERENCES:
- [Derived] Goueffic Y, Della Schiava N, Thaveau F, Rosset E, Favre JP, Salomon du Mont L, Alsac JM, Hassen-Khodja R, Reix T, Allaire E, Ducasse E, Soler R, Guyomarc'h B, Nasr B. Stenting or Surgery for De Novo Common Femoral Artery Stenosis. JACC Cardiovasc Interv. 2017 Jul 10;10(13):1344-1354. doi: 10.1016/j.jcin.2017.03.046. PMID 28683941